CLINICAL TRIAL: NCT00724503
Title: Randomised Comparative Study Of Folfox6m Plus Sir-Spheres® Microspheres Versus Folfox6m Alone As First Line Treatment In Patients With Nonresectable Liver Metastases From Primary Colorectal Carcinoma
Brief Title: FOLFOX Plus SIR-SPHERES MICROSPHERES Versus FOLFOX Alone in Patients With Liver Mets From Primary Colorectal Cancer
Acronym: SIRFLOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STX0206
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Liver Metastases
Keywords: colon cancer; Colorectal carcinoma; liver metastases; SIR-Spheres microspheres; yttrium-90; FOLFOX; bevacizumab; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mFOLFOX6 + SIRT (Experimental): A single injection of SIR-Spheres microspheres into the liver plus systemic chemotherapy consisting of Oxaliplatin + Leucovorin + 5-Fluorouracil (FOLFOX)
  Interventions: Device: SIR-Spheres yttrium-90 microspheres
- mFOLFOX6 (Active Comparator): Systemic chemotherapy consisting of Oxaliplatin + Leucovorin + 5- Fluorouracil (FOLFOX).
  Interventions: Drug: Systemic chemotherapy (FOLFOX)

INTERVENTIONS:
Device: SIR-Spheres yttrium-90 microspheres — SIR-Spheres microspheres (yttrium-90 [Y-90] labelled resin microspheres), hepatic artery injection administered on Day 3 or 4 of cycle 1.
  mFOLFOX6 administered on Day 1 and at the start of each cycle every 14 days: 85 or 60 mg/m2 oxaliplatin by 2-hour intravenous (IV) infusion + 200 mg/m2 leucovorin by 2-hour IV infusion + 400 mg/m2 5-fluorouracil (5-FU) by IV bolus + 2.4 g/m2 5-FU by 46-hour continuous IV infusion.
  Treatment with the biologic agent bevacizumab, if part of standard practice at the participating institution, was permitted at the discretion of the treating Investigator.
  In the event that leucovorin was not available, use of levofolinic acid (the active S enantiomer) was acceptable at half the dose of the racemic leucovorin i.e. 100 mg/m2.
  Other Names: mFOLFOX6m + SIRT; SIR-Spheres Y-90 microspheres
  Arms: mFOLFOX6 + SIRT
Drug: Systemic chemotherapy (FOLFOX) — mFOLFOX6 administered on Day 1 and at the start of each cycle every 14 days: 85 or 60 mg/m2 oxaliplatin by 2-hour intravenous (IV) infusion + 200 mg/m2 leucovorin by 2-hour IV infusion + 400 mg/m2 5-fluorouracil (5-FU) by IV bolus + 2.4 g/m2 5-FU by 46-hour continuous IV infusion.
  Treatment with the biologic agent bevacizumab, if part of standard practice at the participating institution, was permitted at the discretion of the treating Investigator.
  In the event that leucovorin was not available, use of levofolinic acid (the active S enantiomer) was acceptable at half the dose of the racemic leucovorin i.e. 100 mg/m2.
  Other Names: mFOLFOX6
  Arms: mFOLFOX6

SUMMARY:
This study is a randomized multi-center trial that will assess the effect of adding Selective Internal Radiation Therapy (SIRT), using SIR-Spheres microspheres®, to a standard chemotherapy regimen of FOLFOX as first line therapy in patients with non-resectable liver metastases from primary colorectal adenocarcinoma.

Treatment with the biologic agent bevacizumab, if part of the standard of care at participating institutions, is allowed within this study at the discretion of the treating Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal and measurable CT evidence of liver metastases which are not treatable by surgical resection or local ablation.
* Limited extra-hepatic metastases in the lung and/or lymph nodes are permitted (Lung: 5 lesions total, < 1 cm, or 1 single lesion of up to 1.7 cm; Lymph nodules in one single anatomic area (pelvis, abdomen or chest): any number, < 2 cm).
* Suitable for either treatment regimen.
* Prior chemotherapy for metastatic colorectal cancer is not allowed.
* WHO performance status 0-1.
* Adequate hematological, renal and hepatic function.
* Age 18 years or older.
* Willing and able to provide written informed consent.
* Life expectancy of at least 3 months without any active treatment.

Exclusion Criteria

* Evidence of ascites, cirrhosis, portal hypertension, main portal or venous tumor involvement or thrombosis as determined by clinical or radiologic assessment.
* Previous radiotherapy delivered to the upper abdomen.
* Non-malignant disease that would render the patient unsuitable for treatment according to the protocol.
* Peripheral neuropathy > grade 1 (NCI-CTC).
* Dose limiting toxicity with previous adjuvant 5-FU or oxaliplatin chemotherapy.
* Prior non-adjuvant chemotherapy for any malignancy. Adjuvant chemotherapy for colorectal cancer is not an exclusion criteria provided that it was completed more than 6 months before entry into the study.
* Pregnant or breast-feeding.
* Other active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gibbs, MD, Principal Investigator — Melbourne Health; Guy van Hazel, MD, Principal Investigator — Mount Medical Centre
Locations (111):
- United States (21):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - City of Hope Hospital, Duarte, California
  - Florida International University College of Medicine Practice, North Miami Beach, Florida
  - Vanguard Health, Berwyn, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Adventist Hinsdale Hospital, Hinsdale, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Holy Name Hospital, Teaneck, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Altru Health Systems, Grand Forks, North Dakota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St. Mark's Hospital, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin/Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Australia (31):
  - Concord Hospital, Concord, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Nepean Cancer Care Centre, Kingswood, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wesley Medical Centre, Auchenflower, Queensland
  - Cairns Private Hospital, Cairns, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast Health Service District, Southport, Queensland
  - HOCA Gold Coast Centre, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Centre, Ashford, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Queen Elizabeth II Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Bentleigh East, Victoria
  - John Fawkner Private Hospital, Coburg, Victoria
  - Western Hospital, Footscray, Victoria
  - Peninsula Oncology Centre, Frankston, Victoria
  - South Eastern Private, Noble Park, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Ringwood/Knox Private, Ringwood, Victoria
  - Maroondah Public, Ringwood East, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Mount Medical Centre, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (14):
  - OL Vrouw Ziekenhuis Aalst Gastro-Enterologie, Aalst
  - ZNA Middelheim, Antwerp
  - Antwerp University Hospital, Antwerp
  - Imelda Ziekenhuis GI Clinical Research Centre, Bonheiden
  - Sint-Josef Ziekenhuie (Campus Bornem), Bornem
  - Institut Jules Bordet - Centre de Tumeurs d'ULB, Brussels
  - Universiteits Ziekenhuis Gent, Ghent
  - AZ Maria Middelares, Ghent
  - Hospital de Jolimont, Haine-Saint-Paul
  - UZ Leuven, Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - VZW Emmaus St. Maarten Ziekenhuis Mechelen and St. Marten Ziekenhuis Duffel, Mechelen
  - AZ Heilige Familie, Reet
  - Sint-Augustinus Ziekenhuis, Wilrijk
- France (6):
  - CHU de Bordeau, Bordeaux
  - Hospitalier Universitaire de Grenoble C.H.U., La Tronche
  - Centre Hospitalier General de Longjumeau, Longjumeau
  - Hopital de l'Archet II, CHU de Nice, Nice
  - Hospital European Georges Pompidou, Paris
  - Centre Eugene Marquis, Rennes
- Germany (24):
  - Internistische Gemeinschaftspraxis, Altstadt
  - Charite Campus Virchow Klinikum, Berlin
  - Braxiskooperation Bonn, Fachartze fur Innere Medizin, Bonn
  - Johanniterkrankenhaus Bonn, Bonn
  - Universitaetsklinikum Bonn, Bonn
  - Kliniken Essen Mitte, Essen
  - Gemeinschaftspraxis Hamatologie und internistische Onkologie, Essen
  - Universitat Frankfurt Institute fur Diagnostic und Interventionelle Radiologie, Frankfurt
  - Asklepios Klinik Altona, Abt. Radiologie, Neuroradiologie, Nuklearmedizin, Hamburg
  - Universitastsklinikum Saarland, Hamburg
  - Praxisgemeinschaft Dr. med. Peter Sandor und Peter Kohl, Holzkirch
  - Onklogische Praxis Dr. Gerald Gehbauer, Ingolstadt
  - Klinikum Karlsruhe, Stadtisches Klinikum Karlsruhe, Zentralinstitut fur Bildgebende Diagnostik, Karlsruhe
  - Schwerpunktpraxis fur Hamatologie und Onkologie, Magdeburg
  - Klinikum Magdeburg GmbH, Klinik für Hämatologie/Onkologie, Magdeburg
  - Universitaetsklinikum Magdeburg, Magdeburg
  - Universitatsklinikum GieBen und Marburg, Marburg
  - Hamato-Onkologische Schwerpunktspraxis, München
  - Klinikum Bogenhausen, München
  - Klinikum der Universitaet Muenchen, München
  - Klinikum rechts der Isar der TU Munchen, München
  - Schwerpunktspraxis fur Hamatologie und Internistische Onkologie, München
  - Praxis fur Hamatologie und Internnistische Onkologie, Velbert
  - Schwerpunktspraxis und Tagesklinik Dr. Perker/Dr. Sandherr, Weilheim
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare-Zedek Medical Centre, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - TA Sourasky Medical Center, Tel Aviv
- A.O.U. die Bologna, Bologna, Italy
- New Zealand (5):
  - University of Auckland, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Wellington Hospital, Newtown
  - Palmerston North Hospital, Palmerston
- Wojskowy Instytut Medyczny (WIM), Warsaw, Poland
- Spain (2):
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital de Navarra, Servicio de Ongoligia, Planta Baja, Pamplona
- Universitatsspital Zurich, Zurich, Switzerland

REFERENCES:
- [Result] van Hazel GA, Heinemann V, Sharma NK, Findlay MP, Ricke J, Peeters M, Perez D, Robinson BA, Strickland AH, Ferguson T, Rodriguez J, Kroning H, Wolf I, Ganju V, Walpole E, Boucher E, Tichler T, Shacham-Shmueli E, Powell A, Eliadis P, Isaacs R, Price D, Moeslein F, Taieb J, Bower G, Gebski V, Van Buskirk M, Cade DN, Thurston K, Gibbs P. SIRFLOX: Randomized Phase III Trial Comparing First-Line mFOLFOX6 (Plus or Minus Bevacizumab) Versus mFOLFOX6 (Plus or Minus Bevacizumab) Plus Selective Internal Radiation Therapy in Patients With Metastatic Colorectal Cancer. J Clin Oncol. 2016 May 20;34(15):1723-31. doi: 10.1200/JCO.2015.66.1181. Epub 2016 Feb 22. PMID 26903575
- [Derived] Wolstenholme J, Fusco F, Gray AM, Moschandreas J, Virdee PS, Love S, Van Hazel G, Gibbs P, Wasan HS, Sharma RA. Quality of life in the FOXFIRE, SIRFLOX and FOXFIRE-global randomised trials of selective internal radiotherapy for metastatic colorectal cancer. Int J Cancer. 2020 Aug 15;147(4):1078-1085. doi: 10.1002/ijc.32828. Epub 2020 Jan 9. PMID 31840815
- [Derived] Wasan HS, Gibbs P, Sharma NK, Taieb J, Heinemann V, Ricke J, Peeters M, Findlay M, Weaver A, Mills J, Wilson C, Adams R, Francis A, Moschandreas J, Virdee PS, Dutton P, Love S, Gebski V, Gray A; FOXFIRE trial investigators; SIRFLOX trial investigators; FOXFIRE-Global trial investigators; van Hazel G, Sharma RA. First-line selective internal radiotherapy plus chemotherapy versus chemotherapy alone in patients with liver metastases from colorectal cancer (FOXFIRE, SIRFLOX, and FOXFIRE-Global): a combined analysis of three multicentre, randomised, phase 3 trials. Lancet Oncol. 2017 Sep;18(9):1159-1171. doi: 10.1016/S1470-2045(17)30457-6. Epub 2017 Aug 3. PMID 28781171
- [Derived] Virdee PS, Moschandreas J, Gebski V, Love SB, Francis EA, Wasan HS, van Hazel G, Gibbs P, Sharma RA. Protocol for Combined Analysis of FOXFIRE, SIRFLOX, and FOXFIRE-Global Randomized Phase III Trials of Chemotherapy +/- Selective Internal Radiation Therapy as First-Line Treatment for Patients With Metastatic Colorectal Cancer. JMIR Res Protoc. 2017 Mar 28;6(3):e43. doi: 10.2196/resprot.7201. PMID 28351831
- [Derived] Gibbs P, Gebski V, Van Buskirk M, Thurston K, Cade DN, Van Hazel GA; SIRFLOX Study Group. Selective Internal Radiation Therapy (SIRT) with yttrium-90 resin microspheres plus standard systemic chemotherapy regimen of FOLFOX versus FOLFOX alone as first-line treatment of non-resectable liver metastases from colorectal cancer: the SIRFLOX study. BMC Cancer. 2014 Dec 1;14:897. doi: 10.1186/1471-2407-14-897. PMID 25487708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 10 October 2006 and 26 April 2013, 561 patients were screened. 31 screen failures included 2 patients who were randomized twice. 530 patients were randomized in the Intent to treat (ITT) population from 87 centres in Australia, Europe including Belgium, France, Germany, Israel, Italy and Spain, New Zealand and the US.
Groups:
- mFOLFOX6 Plus SIRT: A single injection of SIR-Spheres microspheres into the liver plus systemic chemotherapy consisting of Oxaliplatin + Leucovorin + 5-Fluorouracil (FOLFOX)
- mFOLFOX6 Alone: systemic chemotherapy consisting of Oxaliplatin + Leucovorin + 5-Fluorouracil (FOLFOX)
Period: Overall Study
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
Started | 267 | 263
Completed | 57 | 43
Not Completed | 210 | 220
Not completed — Lost to Follow-up | 4 | 8
Not completed — Withdrawal by Subject | 11 | 23
Not completed — Death | 190 | 182
Not completed — Adverse Event | 1 | 0
Not completed — Not otherwise specified | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone | Total
Number analyzed (Participants) | 267 | 263 | 530
Age, Continuous [Median (Full Range); unit: years] — Population: Age was unknown for 1 patient as patient withdrew consent and records
  years
    number analyzed (Participants) | 267 | 262 | 529
    (all) | 63 [28 to 81] | 63 [23 to 89] | 63 [23 to 89]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was unknown for 1 patient as patient withdrew consent and records
  Participants
    number analyzed (Participants) | 267 | 262 | 529
    Female | 85 | 88 | 173
    Male | 182 | 174 | 356
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 248 | 243 | 491
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 6 | 5 | 11
WHO performance status [Number; unit: participants] — WHO performance status: (0) Able to carry out all normal activity without restriction
  (1) Restricted in physically strenuous activity but ambulatory and able to carry out light work
  participants
    0 | 176 | 175 | 351
    1 | 90 | 87 | 177
    Unknown | 1 | 1 | 2
Primary tumor in situ [Count of Participants; unit: Participants]
  No | 148 | 141 | 289
  Yes | 119 | 121 | 240
  Unknown | 0 | 1 | 1
Extra-hepatic metastases at randomization [Number; unit: participants]
  No | 160 | 159 | 319
  Yes | 107 | 104 | 211
Tumor liver involvement % [Count of Participants; unit: Participants]
  <=25% | 185 | 192 | 377
  >25% | 81 | 70 | 151
  Unknown | 1 | 1 | 2
Synchronous metastases [Count of Participants; unit: Participants] | 241 | 233 | 474

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at Any Site
Description: PFS defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as an increase in the sum of the longest diameters of ≥ 20% and an absolute increase in the sum of the longest diameters of ≥ 5 mm, or the appearance of a new lesion.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
Number analyzed (Participants) | 267 | 263
Months | 10.7 [9.9 to 11.4] | 10.2 [9.4 to 11.3]
Statistical Analysis 1: Comparison: mFOLFOX6 Plus SIRT vs mFOLFOX6 Alone; The null hypothesis tested for the primary efficacy endpoint is rate of progression (months) of SIRT/FOLFOX treatment versus FOLFOX is equal for both groups. The two-sided alternative hypothesis tested with 95% confidence is PFS rate for SIRT/FOLFOX treatment lower to that of FOLFOX; Test type: Superiority; p = 0.551, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.77 to 1.12]

2. Secondary Outcome: Percentage of Participants With Overall Response
Description: Tumour Response Rate per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR) - Disappearance of all target lesions which is confirmed if determined by two observations not less than 4 weeks apart; Partial Response (PR) - >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Through study completion, up to 60 months
Measure: Number; unit: percentage of participants
Groups:
- B: FOLFOX + SIR-Spheres: A single injection of SIR-Spheres microspheres into the liver plus systemic chemotherapy consisting of Oxaliplatin + Leucovorin + 5-Fluorouracil (FOLFOX)
  SIR-Spheres yttrium-90 microspheres: SIR-Spheres microspheres implanted once on the 3rd or 4th day of the first week of the first chemotherapy cycle
  Systemic chemotherapy (FOLFOX): Oxaliplatin 60 mg/m2,IV infusion, q two weeks for first 3 cycles
  Oxaliplatin 85 mg/m2, IV infusion, q two weeks from cycle 4 onwards
  Leucovorin 200 mg/m2, IV infusion, q two weeks
  5-Fluorouracil 400 mg/m2, IV bolus, q two weeks
  5-Fluorouracil 2.4 g/m2, IV infusion, q two weeks
- A: FOLFOX Alone: Systemic chemotherapy consisting of Oxaliplatin + Leucovorin + 5- Fluorouracil (FOLFOX)
  Systemic chemotherapy (FOLFOX): Oxaliplatin 85 mg/m2, IV infusion, q two weeks
  Leucovorin 200 mg/m2, IV infusion, q two weeks
  5-Fluorouracil 400 mg/m2, IV bolus, q two weeks
  5-Fluorouracil 2.4 g/m2, IV infusion, q two weeks
Arm/Group | B: FOLFOX + SIR-Spheres | A: FOLFOX Alone
Number analyzed (Participants) | 267 | 263
percentage of participants | 76.4 | 68.1
Statistical Analysis 1: Comparison: B: FOLFOX + SIR-Spheres vs A: FOLFOX Alone; A sample size of at least 450 patients for the SIRFLOX study was estimated to be needed to detect an increase in the median PFS at any site from 9.4 months to 12.5 months with 80% power and 95% confidence. Taking into account the number of patients who might receive the alternative treatment or lack of imaging data, the sample size was increased to 530. The Null hypothesis is no difference between the treatment arms with respect to PFS; Test type: Superiority; p < 0.05, Log Rank; Hazard Ratio (HR) = 0.75

ADVERSE EVENTS:
Time Frame: From consent until 28 days post last dose of protocol chemotherapy.
Description: Adverse Events monitored for all participants who were randomized and received at least 1 cycle of study treatment.
  Of the 267 in 'mFOLFOX6 Plus SIRT' arm, 18 switched study treatment arms and 3 did not get any treatment. Hence safety population in this arm comprises 246 participants.
  The 'mFOLFOX6 alone' arm includes the initial 263 plus 18 that switched over. 11 did not receive any treatment. Hence safety population in this arm comprises 270 participants.
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
All-Cause Mortality (participants affected / at risk) | 190/246 | 182/270
Serious Adverse Events (participants affected / at risk) | 134/246 | 112/270
Other Adverse Events (participants affected / at risk) | 112/246 | 157/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 Plus SIRT (N=246) | mFOLFOX6 Alone (N=270)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 13 | 4
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Splenic Infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 2 | 2
Angina Pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriospasm Coronary (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 1
Intracardiac Thrombus (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Stress Cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 11 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 2
Anal Inflammation (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 10 | 7
Diarrhoea (Gastrointestinal disorders) | 11 | 8
Duodenal Ulcer (Gastrointestinal disorders) | 3 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 2 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 6 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0
Gastritis Atrophic (Gastrointestinal disorders) | 1 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal Haematoma (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 4 | 6
Intestinal Perforation (Gastrointestinal disorders) | 2 | 3
Large Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 8 | 4
Oesophageal Ulcer (Gastrointestinal disorders) | 1 | 0
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 3 | 2
Rectal Stenosis (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Volvulus Of Small Bowel (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 16 | 3
Asthenia (General disorders) | 3 | 1
Chest Pain (General disorders) | 3 | 0
Chills (General disorders) | 1 | 0
Device Dislocation (General disorders) | 0 | 1
Device Occlusion (General disorders) | 0 | 2
Extravasation (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 0
General Physical Health Deterioration (General disorders) | 1 | 2
Hernia (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0
Infusion Site Pain (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 17 | 12
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 2
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder Perforation (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 3 | 0
Hepatic Fibrosis (Hepatobiliary disorders) | 1 | 0
Hepatic Infarction (Hepatobiliary disorders) | 1 | 0
Hepatic Pain (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 2 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 1
Abdominal Wall Infection (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 1
Acute Sinusitis (Infections and infestations) | 0 | 1
Anorectal Infection (Infections and infestations) | 1 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 0
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 0 | 1
Infusion Site Infection (Infections and infestations) | 1 | 2
Klebsiella Sepsis (Infections and infestations) | 0 | 1
Liver Abscess (Infections and infestations) | 2 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 2 | 2
Neutropenic Sepsis (Infections and infestations) | 1 | 1
Oesophageal Candidiasis (Infections and infestations) | 1 | 0
Pelvic Abscess (Infections and infestations) | 0 | 1
Perihepatic Abscess (Infections and infestations) | 2 | 0
Peritonitis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 4
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Anastomotic Complication (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis Radiation (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Embolisation Syndrome (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Diarrhoea (Injury, poisoning and procedural complications) | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0
Radiation Hepatitis (Injury, poisoning and procedural complications) | 2 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Vascular Procedure Complication (Injury, poisoning and procedural complications) | 1 | 0
Wound Evisceration (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Albumin Decreased (Investigations) | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 3 | 0
Haemoglobin Decreased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 1
Troponin I Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemi (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 4
Hallucination (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Physical Assault (Social circumstances) | 1 | 0
Social Stay Hospitalisation (Social circumstances) | 1 | 0
Abscess Drainage (Surgical and medical procedures) | 0 | 1
Gastrointestinal Surgery (Surgical and medical procedures) | 1 | 0
Hernia Repair (Surgical and medical procedures) | 1 | 0
Surgery NOS (Surgical and medical procedures) | 1 | 0 — NOS: Not Otherwise Specified
Artery Dissection (Vascular disorders) | 1 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 2
Embolism (Vascular disorders) | 1 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 3 | 2
Hypovolaemic Shock (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Peripheral Artery Stenosis (Vascular disorders) | 0 | 1
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0
Peripheral Embolism (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
Venous Thrombosis Limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 Plus SIRT (N=246) | mFOLFOX6 Alone (N=270)
Anaemia (Blood and lymphatic system disorders) | 29 | 38
Febrile Neutropenia (Blood and lymphatic system disorders) | 15 | 5
Leukopenia (Blood and lymphatic system disorders) | 33 | 21
Lymphopenia (Blood and lymphatic system disorders) | 15 | 5
Neutropenia (Blood and lymphatic system disorders) | 66 | 102
Thrombocytopenia (Blood and lymphatic system disorders) | 97 | 47
Abdominal Pain (Gastrointestinal disorders) | 103 | 53
Abdominal Pain Upper (Gastrointestinal disorders) | 77 | 22
Ascites (Gastrointestinal disorders) | 23 | 4
Constipation (Gastrointestinal disorders) | 108 | 91
Diarrhoea (Gastrointestinal disorders) | 103 | 132
Dyspepsia (Gastrointestinal disorders) | 25 | 22
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 18 | 25
Nausea (Gastrointestinal disorders) | 15 | 137
Rectal Haemorrhage (Gastrointestinal disorders) | 23 | 18
Stomatitis (Gastrointestinal disorders) | 45 | 47
Vomiting (Gastrointestinal disorders) | 95 | 74
Asthenia (General disorders) | 39 | 27
Chest Pain (General disorders) | 23 | 10
Fatigue (General disorders) | 26 | 134
Mucosal Inflammation (General disorders) | 40 | 54
Oedema Peripheral (General disorders) | 35 | 17
Pyrexia (General disorders) | 57 | 43
Drug Hypersensitivity (Immune system disorders) | 13 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 15 | 24
Urinary Tract Infection (Infections and infestations) | 19 | 15
Procedural Pain (Injury, poisoning and procedural complications) | 32 | 4
Aspartate Aminotransferase Increased (Investigations) | 13 | 7
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 13 | 8
Neutrophil Count Decreased (Investigations) | 25 | 12
Platelet Count Decreased (Investigations) | 25 | 10
Weight Decreased (Investigations) | 55 | 39
Weight Increased (Investigations) | 15 | 21
White Blood Cell Count Decreased (Investigations) | 15 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 77 | 77
Dehydration (Metabolism and nutrition disorders) | 14 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 32 | 22
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 21 | 16
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 16 | 14
Dizziness (Nervous system disorders) | 25 | 29
Dysgeusia (Nervous system disorders) | 56 | 52
Headache (Nervous system disorders) | 35 | 28
Lethargy (Nervous system disorders) | 13 | 13
Neuropathy Peripheral (Nervous system disorders) | 12 | 15
Paraesthesia (Nervous system disorders) | 32 | 47
Peripheral Sensory Neuropathy (Nervous system disorders) | 41 | 43
Polyneuropathy (Nervous system disorders) | 13 | 17
Anxiety (Psychiatric disorders) | 9 | 15
Depression (Psychiatric disorders) | 15 | 8
Insomnia (Psychiatric disorders) | 35 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 61 | 68
Hiccups (Respiratory, thoracic and mediastinal disorders) | 13 | 15
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 29 | 31
Dry Skin (Skin and subcutaneous tissue disorders) | 20 | 19
Palmar-Plantar Erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 21 | 27
Rash (Skin and subcutaneous tissue disorders) | 32 | 35
Hypertension (Vascular disorders) | 42 | 48
Hypotension (Vascular disorders) | 13 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No